CLINICAL TRIAL: NCT00985777
Title: A Phase I Dose-Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Vitamin E δ-Tocotrienol Administered to Subjects With Resectable Pancreatic Exocrine Neoplasia
Brief Title: Vitamin E δ-Tocotrienol Administered to Subjects With Resectable Pancreatic Exocrine Neoplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15630; 1R01CA129227-01A1 (NIH)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Pancreatic Neoplasms
Keywords: pancreas; resectable; pancreatic tumor; pancreatic ductal adenocarcinoma; intraductal papillary mucinous neoplasm of the pancreas; mucinous cystic neoplasm; pancreatic exocrine neoplasia
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Intraductal Neoplasms | interventions — tocotrienol, delta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I Dose Escalation (Experimental): Vitamin E δ-Tocotrienol will be administered orally as a single agent twice daily for 14 consecutive days and one dose on Day 15.
  Interventions: Drug: Vitamin E δ-Tocotrienol

INTERVENTIONS:
Drug: Vitamin E δ-Tocotrienol — Vitamin E δ-Tocotrienol is supplied as 100-mg, 200-mg, and 400-mg capsules. The investigator (or designee) will have records of the number of participants treated within a specific cohort and will determine which treatment cohort to assign newly enrolled participants.
  Other Names: Delta-tocotrienol

SUMMARY:
The purpose of this study is to determine the safest dose of the study drug Vitamin E Delta-tocotrienol, how often it should be taken, and how well people with pancreatic tumors tolerate Vitamin E Delta-tocotrienol.

DETAILED DESCRIPTION:
Delta-tocotrienol is a natural Vitamin E compound that has been consumed by humans as a dietary supplement. The Food and Drug Administration (FDA) has not approved it for sale as a drug. Vitamin E Delta-tocotrienol is being investigated for the prevention and treatment of pancreatic tumors. The usefulness of the Vitamin E Delta-tocotrienol in treating human tumors is unknown.

This study consists of the following: (1) a Pre-Treatment Period in which participants are consented and qualified for the study; (2) a Study Treatment Period in which participant will receive Vitamin E δ-Tocotrienol administered orally twice daily for 14 (±2) consecutive days and once on the day of surgery, with associated pharmacokinetic and pharmacodynamic sampling; (3) a Post Treatment Period in which laboratory and physical examinations are performed. Adverse events will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a resectable tumor or cyst arising from the pancreatic exocrine gland (pancreatic ductal adenocarcinoma, intraductal papillary mucinous neoplasm of the pancreas, or mucinous cystic neoplasm of the pancreas) and is undergoing surgical resection of the neoplasm.
* The patient is not a candidate for neoadjuvant chemoradiation therapy (i.e., patients with borderline resectable pancreatic ductal adenocarcinoma who are known to benefit from neoadjuvant treatment regimens).
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* The patient has adequate organ function as follows: Serum creatinine ≤1.5 mg/dL or calculated creatinine clearance >60 mL/min; Bilirubin ≤ the institutional upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal if no liver involvement or ≤5 times the upper limit of normal with liver involvement; absolute neutrophil count (ANC) ≥ 1000mm³; Platelet count ≥100,000/mm³.
* The patient has the capability of understanding the informed consent document and has signed the informed consent document.
* Sexually active patients (male and female) must use medically acceptable methods of contraception during the course of the study.
* Female patients of childbearing potential must have a negative pregnancy test at screening.
* Able to understand and comply with the requirements of the protocol.

Exclusion Criteria:

* The patient is receiving concomitant radiotherapy, chemotherapy, other antineoplastic therapy, or investigational therapy (other than the investigational therapy under study).
* The patient has received radiation therapy, chemotherapy, other anti-neoplastic therapy, or investigational therapy within 30 days prior to first dose of study drug.
* The patient has had prior major surgery within 30 days prior to first dose of study drug.
* The patient has active infection or fever >38.5 C within 3 days prior to first dose of study drug.
* The patient has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* The patient is unable or unwilling to stop taking vitamins, herbal remedies, or nonprescription medications.
* The patient is pregnant or breastfeeding.
* The patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
* The patient is a candidate for neo-adjuvant radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-09; Primary Completion 2015-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 12 weeks per participant
  To determine the recommended Phase II dose of Vitamin E δ-Tocotrienol which will be defined as the biologic effective dose (BED) which induces significant apoptosis in the pancreatic neoplastic cells of resected tumor specimens following oral administration of Vitamin E δ-Tocotrienol twice daily for 14 (± 2)days prior to surgery, and one dose the day of surgery.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | 12 weeks per participant
  To characterize the safety and tolerability of Vitamin E δ-Tocotrienol when orally administered at up to 5.6 times the predicted biological effective dose (1600mg twice daily) for 14 (± 2) consecutive days and one dose the day of surgery in patients with pancreatic neoplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Springett, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Springett GM, Husain K, Neuger A, Centeno B, Chen DT, Hutchinson TZ, Lush RM, Sebti S, Malafa MP. A Phase I Safety, Pharmacokinetic, and Pharmacodynamic Presurgical Trial of Vitamin E delta-tocotrienol in Patients with Pancreatic Ductal Neoplasia. EBioMedicine. 2015 Nov 14;2(12):1987-95. doi: 10.1016/j.ebiom.2015.11.025. eCollection 2015 Dec. PMID 26844278